CLINICAL TRIAL: NCT02760316
Title: A Phase I, Randomised, Single-blind Study to Asses the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of AZD9567 in Healthy Volunteers Using Prednisolone as Positive Control
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of AZD9567.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6470C00002
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Healthy Volunteers; Obese; Insulin Resistant Subjects; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Obesity | interventions — AZD9567; Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- AZD9567 oral suspension of 10 mg (Experimental): Participants will receive oral supension of 10 mg dose strength
  Interventions: Drug: AZD9567 10 mg
- AZD9567 oral suspension of 20 mg (Experimental): Participants will receive oral suspension of 20 mg dose strength
  Interventions: Drug: AZD9567 20 mg
- AZD9567 oral suspension of 40 mg (Experimental): Participants will receive oral suspension of 40 mg dose strength
  Interventions: Drug: AZD9567 40 mg
- AZD9567 oral suspension of 80 mg (Experimental): Participants will receive oral suspension of 80mg dose strength
  Interventions: Drug: AZD9567 80 mg
- Prednisolone oral capsules of 20 mg (Active Comparator): Participants will receive oral capsules of 5 mg dose strength
  Interventions: Drug: Prednisolone 20 mg
- AZD9567 oral suspension of 125 mg (Experimental): Participants will receive oral suspension of 125 mg dose strength
  Interventions: Drug: AZD9567 125 mg
- AZD9567 oral suspension of 155 mg (Experimental): Participants will receive oral suspension of 155 mg dose strength
  Interventions: Drug: AZD9567 155 mg
- Prednisolone oral capsules of 5 mg (Active Comparator): Participants will receive oral capsules of 5 mg dose strength
  Interventions: Drug: Prednisolone 5 mg
- Prednisolone oral capsules of 40 mg (Active Comparator): Participants will receive oral capsules of 5 mg dose strength
  Interventions: Drug: Prednisolone 40 mg

INTERVENTIONS:
Drug: AZD9567 10 mg — Oral suspension Multiple doses 5 days of treatment Once daily
  Arms: AZD9567 oral suspension of 10 mg
Drug: AZD9567 20 mg — Oral suspension Multiple doses 5 days of treatment Once daily
  Arms: AZD9567 oral suspension of 20 mg
Drug: AZD9567 40 mg — Oral suspension Multiple doses 5 days of treatment Once daily
  Arms: AZD9567 oral suspension of 40 mg
Drug: AZD9567 80 mg — Oral suspension Multiple doses 5 days of treatment Once daily
  Arms: AZD9567 oral suspension of 80 mg
Drug: Prednisolone 20 mg — Oral Multiple doses 5 days of treatment Once daily
  Arms: Prednisolone oral capsules of 20 mg
Drug: AZD9567 125 mg — Oral Multiple doses 5 days of treatment Once daily
  Arms: AZD9567 oral suspension of 125 mg
Drug: AZD9567 155 mg — Oral Multiple doses 5 days of treatment Once daily
  Arms: AZD9567 oral suspension of 155 mg
Drug: Prednisolone 5 mg — Oral Multiple doses 5 days of treatment Once daily
  Arms: Prednisolone oral capsules of 5 mg
Drug: Prednisolone 40 mg — Oral Multiple doses 5 days of treatment Once daily
  Arms: Prednisolone oral capsules of 40 mg

SUMMARY:
A study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of AZD9567.

DETAILED DESCRIPTION:
This is a phase 1, randomised, single-blind, multiple ascending dose, double-dummy sequential group study in healthy subjects .

The study is planned to have 6 cohorts with the option to include up to two additional cohorts if deemed necessary. Nine subjects participated in the first cohort (7 subjects randomised to receive AZD9567 and 2 subjects randomised to receive prednisolone 20 mg)and eleven subjects will participate in subsequent 3 cohorts (7 subjects will be randomised to receive AZD9567 and 4 subjects randomised to receive prednisolone 20 mg). A cohort 5 was included in the study in version 4.0 of the CSP. In this cohort two doses of prednisolone was tested, 5 mg and 20 mg. Up to six dose levels of AZD9567 are planned to be tested in the study and an additional cohort will be used in case any previous dose needs to be repeated or a new lower dose explored (ref CSP 5.0).

Therefore a maximum of 95 individuals could be included in the study (as stated in version 5.0 of this protocol). Subjects will be dosed for 5 consecutive days and a follow-up visit will occur 10-14 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-childbearing potential female subject, aged 18 to 55 years (both inclusive) with suitable veins for cannulation or repeated venipuncture. Explanatory note: Female subjects must be of non-childbearing potential, confirmed at screening by fulfilling study predefined criteria
2. Body mass index (BMI) between 18 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
3. Serum cortisol levels within normal limits at Screening (collected as part of the clinical chemistry panel) at the discretion of the Investigator.
4. Able to understand, read and speak the language of the ICD approved by the EC/IRB
5. Provision of signed and dated, written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. History of any clinically important disorder which, in opinion of the Investigator, may either put the subject at risk or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. History or presence of dyspepsia or oral intolerance to steroids.
4. History of or active or latent tuberculosis (TB), or at risk for having acquired TB (social workers or prison staff in countries with endemic rates of TB, having lived with patients with known TB).
5. History suggesting abnormal immune function, as judged by the Investigator.
6. History of severe affective disorder including depressive or maniac-depressive illness.
7. History of previous steroid psychosis
8. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
9. Any latent or chronic infections or at risk of infection, or history of skin abscesses within 90 days prior to the first administration of IMP at the discretion of the Investigator.
10. Any clinically important laboratory abnormalities (serum biochemistry, hematology, coagulation or urinalysis results) at Screening or prior to randomisation, as judged by the Investigator. Explanatory note: In particular a subject with an abnormal value (2x upper level of normal) for alkaline phosphatase (ALP), alanine aminotransferase (ALT) or aspartate aminotransferase (AST), serum creatinine (1.2x upper level of normal), and/or above the upper level of normal in serum bilirubin, or with an abnormal value for haemoglobin (Hb), white blood cell (WBC) and/or absolute neutrophil count below the normal limit will be excluded.
11. Any positive result at Screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and/or human immunodeficiency virus (HIV).
12. Abnormal vital signs after 10 minutes supine rest.

    Explanatory note: Deviations from normal vital signs within the following ranges will not be allowed as any of the following:
    * Systolic BP (SBP) < 90mmHg or > 140 mmHg
    * Diastolic BP (DBP) < 50mmHg or > 90 mmHg
    * Heart rate < 50 or > 90 beats per minute (bpm)
13. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and 12-lead ECG that may interfere with the interpretation of QTc changes Explanatory note: this also includes abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
14. Prolonged QTcF > 450 ms or family history of long QT syndrome.
15. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
16. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation.
17. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms.

    Explanatory note: Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation.
18. Known or suspected history of drug abuse in the last 6 months, as judged by the Investigator.
19. Smokers that smoke ≥ 5 cigarettes/pipes per day, or use tobacco in any other form. Smoking will not be allowed during the study treatment period (Day -2 to Day 6) (1 e-cigarette = 1 cigarette).
20. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
21. Positive screen for drugs of abuse or alcohol at Screening or on admission to the clinical unit.
22. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity to drugs with a similar chemical structure or class to study drugs.
23. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the Investigator.
24. Receipt of live or live attenuated vaccine within 4 weeks prior to the first administration of IMP.
25. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
26. Use of any prescribed or non-prescribed medication during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life. Explanatory note: the prohibited medication includes antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals
27. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
28. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months or 5 half-lifes, whatever is the longest of the first administration of IMP.

    Explanatory note: the period of exclusion begins three months after the final dose or one month after the last visit whichever is the longest. Subjects consented and screened, but not randomised in this study or a previous phase I study, are not excluded.
29. Vulnerable subject, e.g., kept in detention, protected adult under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
30. Involvement of any Astra Zeneca or PAREXEL or study site employee or their close relatives.
31. Judgment by the Investigator that the subject should not participate in the study Explanatory note: for example, if the subject has any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data, or is considered unlikely to comply with study procedures, restrictions and requirements, the subject should not be randomised.
32. Subject who is a vegan or has medical dietary restrictions.
33. Subject who cannot communicate reliably with the Investigator/site staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events (AEs) | Up to 5 days
  Adverse events will be summarized by each dose of AZD9567, pooled prednisolone 20 mg and pooled AZD9567 doses. Tabulations will include causality and severity (mild, moderate and severe), where applicable, and be presented by System Organ Class (SOC) and Preferred Term (PT) where applicable.
Safety and tolerability: Vital signs (blood pressure [BP], pulse rate, weight and oral body temperature) | Up to 5 days
  Descriptive statistics will be presented by treatment and time point for both observed values and changes from baseline, based on the safety analysis sets. The incidence of clinically notable vital sign abnormalities (vital signs outside the predefined criteria) will be summarized.
Safety and tolerability: Clinical laboratory safety evaluations (hematology, serum biochemistry [including S-cortisol and basal S-DHEAS], coagulation and urinalysis) | Up to 5 days
  Summary tabulations will be presented by treatment including observed values and changes from baseline.
  Shift tables will be presented to show the shifts from baseline to the minimum and maximum post-baseline measurements, respectively, by treatment, based on the safety analysis set.
Safety and tolerability: Electrocardiograms (12-lead dECGs, safety ECG's, and telemetry) | Up to 5 days
  Results of the safety ECGs, including normal/abnormal and specific findings will be listed for each subject.
Safety and tolerability: Physical examinations | Up to 5 days
  The results of the physical examination will be listed by body system for each subject.

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Observed maximum concentration (Cmax) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Area Under the curve from 0 to last quantifiable (AUC (0-last)) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Area Under the curve from 0 to 24h (AUC (0-24)) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Area Under the curve from 0 to infinity (AUC(0-inf)) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Area Under the curve from 0 to last quantifiable divided by the dose (AUC(0-last)/D) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Area Under the curve from 0 to 24h divided by the dose (AUC(0-24)/D) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Area Under the curve from 0 to infinity divided by the dose (AUC/D) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Observed maximum concentration divided by the dose (Cmax/D) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Time to reach maximum concentration (tmax) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Terminal rate constant (λz) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Terminal half-life (t1/2) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Apparent clearance divided by AUC (CL/F) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Aparent volume of distribution estimated by dividing de apparent clearance (Vz/F) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: Average plasma concentration (Cav) | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacokinetic parameter: fluctuation index | Up to 5 days
  Plasma concentrations, and plasma PK parameters will be summarized by dose level of AZD9567 using descriptive statistics (n, geometric mean, geometric coefficient of variation [CV%], arithmetic mean, arithmetic Standard Deviation (SD), minimum, median and maximum) based on the respective PK analysis sets.
Pharmacodynamic parameter: Plasma glucose measured by Oral Glucose Tolerance Test (OGTT) | Up to 5 days
  Concentration data for the OGTT (plasma glucose) will be listed and summarized by treatment, visit and time point. Each of the plasma glucose AUC (total net and incremental) parameters (0 to 2 hours and 0 to 4 hours) will be listed and summarized (including changes from baseline for the AUC values, where the baseline is the AUC values measured on Day -1) by visit and treatment for the final clinical study report. In addition, the glucose ratio values by time point and their corresponding AUCs will also be summarized.
Pharmacodynamic parameter: Serum insulin measured by Oral Glucose Tolerance Test (OGTT) | Up to 5 days
  Concentration data for the OGTT (serum insulin) will be listed and summarized by treatment, visit and time point. Each of the serum insulin AUC (total net and incremental) parameters (0 to 2 hours and 0 to 4 hours) will be listed and summarized (including changes from baseline for the AUC values, where the baseline is the AUC values measured on Day -1) by visit and treatment for the final clinical study report. In addition, the serum insulin ratio values by time point and their corresponding AUCs will also be summarized.
Pharmacodynamic parameter: Serum C-peptide measured by Oral Glucose Tolerance Test (OGTT) | Up to 5 days
  Concentration data for the OGTT (serum C-peptide) will be listed and summarized by treatment, visit and time point. Each of the serum C-peptide AUC (total net and incremental) parameters (0 to 2 hours and 0 to 4 hours) will be listed and summarized (including changes from baseline for the AUC values, where the baseline is the AUC values measured on Day -1) by visit and treatment for the final clinical study report.

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL Early Phase Clinical Unit, Berlin; Pablo ForteSoto, Dr., Principal Investigator — PAREXEL Early Phase Clinical Unit, London
Locations (2):
- Research Site, Berlin, Germany
- Research Site, Harrow, United Kingdom

REFERENCES:
- [Derived] Hegelund Myrback T, Prothon S, Edman K, Leander J, Hashemi M, Dearman M, Edenro G, Svanberg P, Andersson EM, Almquist J, Ammala C, Hendrickx R, Taib Z, Johansson KA, Berggren AR, Keen CM, Eriksson UG, Fuhr R, Carlsson BCL. Effects of a selective glucocorticoid receptor modulator (AZD9567) versus prednisolone in healthy volunteers: two phase 1, single-blind, randomised controlled trials. Lancet Rheumatol. 2020 Jan;2(1):e31-e41. doi: 10.1016/S2665-9913(19)30103-1. Epub 2019 Dec 9. PMID 38258274